CLINICAL TRIAL: NCT06840977
Title: RETROSPECTIVE OBSERVATIONAL STUDY OF CHEMOTHERAPY IN ELDERLY PATIENTS IN THE FIRST-LINE TREATMENT OF METASTATIC COLORECTAL CANCER
Brief Title: COLON ERDERLY LOW DOSE
Acronym: CELOW
Status: Not yet recruiting | Type: Observational
Sponsor: Matteo Clavarezza (Other)
Responsible Party: Sponsor-Investigator, Matteo Clavarezza, MD, Ente Ospedaliero Ospedali Galliera
Organization: Ente Ospedaliero Ospedali Galliera (Other)
Other Study IDs: CELOW
Record Dates: First submitted 2025-02-18; First posted 2025-02-21 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Colon Adenocarcinoma
Keywords: metastatic colorectal adenocarcinom; low doses; chemotherapy; monoclonal antibodies
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Retrospective: PATIENTS AGED 70 YEARS AND OVER IN FIRST-LINE TREATMENT OF METASTATIC COLORECTAL CANCER

SUMMARY:
In this retrospective observational study, the case series of patients undergoing first-line treatment for metastatic colorectal adenocarcinoma with doublet fixed-dose and reduced-dose chemotherapy in combination with full-dose monoclonal antibody in patients aged 70 years or older is collected.

DETAILED DESCRIPTION:
Treatment in the elderly first-line patient of metastatic colorectal cancer is often conditioned by the age and general condition of the patient.

Such treatment involves the combination of chemotherapy and biological therapy targeted on the basis of the site and genetic mutations of the colorectal tumour, in particular RAS and BRAF.

With regard to targeted biologic therapy, the choice of monoclonal antibody is determined by tumour site and mutations. In particular, for right-sided and/or RAS/BRAF mutated tumours anti-VEGF therapy with Bevacizumab is the best option, whereas for left-sided and RAS/BRAF WT tumours monoclonal antibodies Panitumunab or Cetuximab are the choice.

In the elderly patient, the intensity of chemotherapy to be combined with targeted biologic therapy varies according to the patient's age, general condition and treatment goals. In particular for patients aged 70 years or older, a valid option is the combination of monochemotherapy with fluorodrugs in combination with bevacizumab. In addition, an Italian randomised trial tested monochemotherapy with 5-Fluorouracil in combination with Panitumumab in RAS WT/BRAF WT tumours and obtained the same efficacy as a doublet of chemotherapy with FOLFOX also in combination with Panitumumab.

Full-dose doublet chemotherapy is hardly feasible in the elderly patient because of the frailty of these patients and the high risk of toxicity.

In this retrospective observational study, we report on the case series of patients undergoing first-line treatment for metastatic colorectal adenocarcinoma with doublet of fixed-dose and reduced-dose chemotherapy in combination with full-dose monoclonal antibody in patients 70 years of age and older.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with metastatic colorectal adenocarcinoma not treated with any therapy in the metastatic phase. Previous (neo)-adjuvant treatment with fluoroderivatives with or without Oxaliplatin is permitted.
2. Age ≥ 70 years
3. G8 score ≥ 12
4. Patients with colorectal adenocarcinoma MSS
5. Patients with BRAF WT colorectal adenocarcinoma
6. Ability to understand and sign the informed consent form.

Exclusion Criteria:

1. Patients with MSI tumours
2. Patients with BRAF V600E mutated tumours
3. Patients not eligible for doublet chemotherapy by clinical decision

Ages: 70 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The study population includes patients aged 70 years and older, with metastatic colorectal adenocarcinoma, MSS, BRAF WT, with a G8 score greater than or equal to 12, candidates for metastatic first-line treatment
Sampling Method: Probability Sample
Enrollment: 51 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Neutropenia incidence | 24 months
  overall incidence of grade 4 neutropenia or febrile neutropenia of less than 8%
Diarrehea incidence | 24 months
  incidence of grade 3-4 diarrhea of less than 8%.

SECONDARY OUTCOMES:
PFS | 24 months
  Progression Free Survival (PFS), i.e. the time from day 1 of cycle 1 of treatment to the date of progression or death, whichever occurs first
OS | 24 months
  Overall Survival (OS), which is the time between the date of cycle day 1 of treatment and death
differences in toxicity of anti-VEGF monoclonal antibodies | 24 months
  Assess toxicity between in ANTI-VEGF monoclonal antibodies
differences in toxicity of anti-EGFR monoclonal antibodies | 24 months
  Assess toxicity between in ANTI-EGFR monoclonal antibodies

CONTACTS AND LOCATIONS:
Overall Officials: Matteo Clavarezza, Principal Investigator — E.O. Ospedali Galliera
Locations (1):
- E.O. Ospedali Galliera, Genoa, Liguria, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Stueger A, Joerger M, De Nys K. Geriatric evaluation methods in oncology and their use in clinical studies: A systematic literature review. J Geriatr Oncol. 2024 Apr;15(3):101684. doi: 10.1016/j.jgo.2023.101684. Epub 2023 Dec 9. PMID 38072709
- [Result] Takashima A, Hamaguchi T, Mizusawa J, Nagashima F, Ando M, Ojima H, Denda T, Watanabe J, Shinozaki K, Baba H, Asayama M, Hasegawa S, Masuishi T, Nakata K, Tsukamoto S, Katayama H, Nakamura K, Fukuda H, Kanemitsu Y, Shimada Y; Colorectal Cancer Study Group in Japan Clinical Oncology Group (JCOG). Oxaliplatin Added to Fluoropyrimidine/Bevacizumab as Initial Therapy for Unresectable Metastatic Colorectal Cancer in Older Patients: A Multicenter, Randomized, Open-Label Phase III Trial (JCOG1018). J Clin Oncol. 2024 Nov 20;42(33):3967-3976. doi: 10.1200/JCO.23.02722. Epub 2024 Aug 26. PMID 39186709
- [Result] Lonardi S, Rasola C, Lobefaro R, Rossini D, Formica V, Scartozzi M, Frassineti GL, Boscolo G, Cinieri S, Di Donato S, Pella N, Bergamo F, Raimondi A, Arnoldi E, Antonuzzo L, Granetto C, Zustovich F, Ronzoni M, Leo S, Morano F, Loupakis F, Buggin F, Zagonel V, Fassan M, Cremolini C, Boni L, Pietrantonio F; GONO Foundation Investigators. Initial Panitumumab Plus Fluorouracil, Leucovorin, and Oxaliplatin or Plus Fluorouracil and Leucovorin in Elderly Patients With RAS and BRAF Wild-Type Metastatic Colorectal Cancer: The PANDA Trial by the GONO Foundation. J Clin Oncol. 2023 Dec 1;41(34):5263-5273. doi: 10.1200/JCO.23.00506. Epub 2023 Aug 3. PMID 37535876
- [Result] Cunningham D, Lang I, Marcuello E, Lorusso V, Ocvirk J, Shin DB, Jonker D, Osborne S, Andre N, Waterkamp D, Saunders MP; AVEX study investigators. Bevacizumab plus capecitabine versus capecitabine alone in elderly patients with previously untreated metastatic colorectal cancer (AVEX): an open-label, randomised phase 3 trial. Lancet Oncol. 2013 Oct;14(11):1077-1085. doi: 10.1016/S1470-2045(13)70154-2. Epub 2013 Sep 10. PMID 24028813
- [Result] Yoshino T, Cervantes A, Bando H, Martinelli E, Oki E, Xu RH, Mulansari NA, Govind Babu K, Lee MA, Tan CK, Cornelio G, Chong DQ, Chen LT, Tanasanvimon S, Prasongsook N, Yeh KH, Chua C, Sacdalan MD, Sow Jenson WJ, Kim ST, Chacko RT, Syaiful RA, Zhang SZ, Curigliano G, Mishima S, Nakamura Y, Ebi H, Sunakawa Y, Takahashi M, Baba E, Peters S, Ishioka C, Pentheroudakis G. Pan-Asian adapted ESMO Clinical Practice Guidelines for the diagnosis, treatment and follow-up of patients with metastatic colorectal cancer. ESMO Open. 2023 Jun;8(3):101558. doi: 10.1016/j.esmoop.2023.101558. Epub 2023 May 24. PMID 37236086
- See also: CTCAE criteria v5 — https://ctep.cancer.gov/protocoldevelopment/electronic_applications/docs/ctcae_v5_quick_reference_5x7.pdf